CLINICAL TRIAL: NCT05942183
Title: The Relationship Between Optic Nerve Sheath Diameter and Postoperative Delirium in Open Heart Surgery
Brief Title: Optic Nerve Sheath Diameter is Associated With Postoperative Delirium in Patients Undergoing Open Heart Surgery
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, Aynur Kaynar, principle investigator, Samsun University
Other Study IDs: SÜKAEK-2023 11/7
Record Dates: First submitted 2023-06-13; First posted 2023-07-12 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Delirium, Postoperative; Cardiac Disease; Cardiac Valve Disease
Keywords: optic nerve sheath diameter; cardiac surgery; ultrasound
MeSH Terms: conditions — Emergence Delirium; Heart Diseases; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CAM-ICU positive: delirium positive
  Interventions: Diagnostic Test: ONSD
- CAM-ICU negative: delirium negative
  Interventions: Diagnostic Test: ONSD

INTERVENTIONS:
Diagnostic Test: ONSD — ultrasound measurement of the optic nerve sheath diameter

SUMMARY:
Although the incidence of delirium after cardiac surgery is high, it is not sufficiently recognized. The long-term effects of delirium are likely to be underestimated. In this study, the investigators aimed to examine the relationship between optic nerve sheath diameter and postoperative delirium in open hearth surgery.

DETAILED DESCRIPTION:
Postoperative delirium is characterized by widespread brain involvement and its incidence is between 6% and 30%. It appears twice as often after cardiac and vascular surgery than other types of surgery. The correlation between optic nerve sheath diameter (ONSD) and invasive intracranial pressure measurement is excellent. ONSD reduction has the potential to indicate intracranial hypoperfusion causing delirium. In this observational study, patients aged 18 years and over who will undergo open heart surgery will be examined. ONSD will be measured using ultrasound five times in the perioperative period (t0: pre-induction, t1: post-induction, t2: onset of cardiopulmonary bypass (CPB), t3: post-CPB, and t4: post-ICU admission). The Confusion Assessment Method for the ICU (CAM-ICU) test will be used to examine delirium in the ICU. Whether the change in ONSD is an independent risk factor for delirium will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 year old
* Elective open heart surgery

Exclusion Criteria:

* psychiatric illness
* neurological disease
* ophthalmic disease
* previous eye surgery
* perioperative cerebrovascular disease
* need for postoperative intraaortic balloon or extracorporeal support system

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who will undergo elective open heart surgery will be included in the study.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
The relationship between ONSD and postoperative delirium in cardiac surgery | 6 months
  Peroperatively measured ONSD will be compared with the development of postoperative delirium.
Incidence of delirium after open heart surgery | 6 months
  Using the CAM-ICU test for delirium definition

CONTACTS AND LOCATIONS:
Locations (1):
- Aynur Kaynar, Samsun, Turkey (Türkiye)

REFERENCES:
- [Background] Heyer EJ, DeLaPaz R, Halazun HJ, Rampersad A, Sciacca R, Zurica J, Benvenisty AI, Quest DO, Todd GJ, Lavine S, Solomon RA, Connolly ES Jr. Neuropsychological dysfunction in the absence of structural evidence for cerebral ischemia after uncomplicated carotid endarterectomy. Neurosurgery. 2006 Mar;58(3):474-80; discussion 474-80. doi: 10.1227/01.NEU.0000197123.09972.EA. PMID 16528187
- [Background] Smith W, Whitlock EL. Cardiac surgery, ICU sedation, and delirium: is dexmedetomidine the silver bullet? Curr Opin Anaesthesiol. 2023 Feb 1;36(1):50-56. doi: 10.1097/ACO.0000000000001207. Epub 2022 Nov 7. PMID 36342329
- [Background] Zhang X, Medow JE, Iskandar BJ, Wang F, Shokoueinejad M, Koueik J, Webster JG. Invasive and noninvasive means of measuring intracranial pressure: a review. Physiol Meas. 2017 Jul 24;38(8):R143-R182. doi: 10.1088/1361-6579/aa7256. PMID 28489610
- [Background] Sekhon MS, Griesdale DE, Robba C, McGlashan N, Needham E, Walland K, Shook AC, Smielewski P, Czosnyka M, Gupta AK, Menon DK. Optic nerve sheath diameter on computed tomography is correlated with simultaneously measured intracranial pressure in patients with severe traumatic brain injury. Intensive Care Med. 2014 Sep;40(9):1267-74. doi: 10.1007/s00134-014-3392-7. Epub 2014 Jul 18. PMID 25034476
- [Derived] Kaynar A, Komurcu O, Bahsi E, Aydin AO, Karal IH, Akyurt D, Tulgar S, Suren M. Optic nerve sheath diameter is associated with postoperative delirium in patients undergoing open heart surgery. BMC Anesthesiol. 2025 Jul 1;25(1):309. doi: 10.1186/s12871-025-03194-9. PMID 40596877